CLINICAL TRIAL: NCT00391261
Title: A Prospective Open-label Trial of Metformin for Weight Control of Pediatric Patients on Atypical Antipsychotic Medications.
Brief Title: An Open-label Trial of Metformin for Weight Control of Pediatric Patients on Antipsychotic Medications.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: American Psychiatric Association (Other)
Responsible Party: Jean Frazier, MD, Cambridge Health Alliance
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-0143/12/05
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2008-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Bipolar Disorder; Autism Spectrum Disorders
Keywords: weight gain; obesity; metabolism
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Autism Spectrum Disorder; Weight Gain; Obesity | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Metformin — open-label, flexible dosing
  Other Names: Glucophage

SUMMARY:
The aim of this study is to evaluate the effectiveness, safety, and tolerability of metformin treatment in children and adolescents suffering from weight gain secondary to use of atypical antipsychotic medications. In this 12 week, open-label study we will investigate metformin's effects on weight control and/or weight loss. We hypothesize that metformin would prevent further weight gain or lead to weight loss, resulting in amelioration of one of the most significant side effects of atypical antipsychotic use.

DETAILED DESCRIPTION:
Patients taking olanzapine, risperidone, or quetiapine with increased BMI of at least 10% over the previous 2 months of atypical therapy will be eligible for the study. Subjects will need to have been on a stable dose of their antipsychotic medications at the time of enrollment (stable x2 weeks) and will remain on the same atypical dose, if possible, throughout the study. The dosing of metformin will start at 500mg per day and increase up to a maximum dose of 1500mg daily. Determination of weight gain during the course of the study will be based on the subject's weight at enrollment and subsequent visits. The patients will be asked not to vary their dietary or physical activity habits during the study.

Interpretation of Data: The study's primary outcome measure will be change in weight and body mass index at 12 weeks of metformin treatment. Additionally, skin-fold test and abdominal girth will be measured at baseline and endpoint.

Risks: Generally, metformin is well-tolerated. However, there may be unknown risks associated with exposure to a new medication in a clinical population where this specific compound has not been studied extensively. The general and rare side effects are listed below. These risks will be minimized by careful monitoring and higher than standard of care safety evaluations. In addition, an individual's symptoms could potentially remain unchanged or worsen by initiating this medication, or from delaying initiation of a potentially more effective alternative treatment. For these reasons, participation in the study is entirely voluntary and consent may be withdrawn at any time without any repercussions and will result in the patient being immediately discontinued from the study. If at any time the clinician believes that the patient is not benefiting from the study, the study will be discontinued and endpoint measures will be obtained if possible. A risk-benefit analysis, weighing clinical improvement against side effects will be done at each visit and will determine further inclusion in the study.

Subjects and their guardians will be asked repeatedly to inform study staff of any side effects. Subjects are informed of the potential side effects and the importance of alerting study staff to the side effects in the consent and assent forms. Side effect data will be collected at baseline and every other week, but subjects are encouraged to give relevant information at every clinical evaluation.

Alternative treatments include no treatment with an attendant risk of increased weight gain, potentially leading to health hazard. Other medications that are available are not extensively used and widely accepted. These other medication options will be discussed as alternatives during the consent process. Also, life-style modifications including healthy diet habits and increased physical activity will be discussed during the consent process as well.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 10-18 years.
2. A DSM-IV diagnosis of bipolar disorder schizophrenia spectrum disorder, or pervasive developmental disorder.
3. Ability to give assent.
4. At least 10% increase in body mass index (BMI) within the past 2 months of quetiapine, olanzapine, or risperidone treatment, per parent or physician report.
5. On stable dose of quetiapine, olanzapine, or risperidone x2 weeks.
6. Otherwise medically stable.

Exclusion Criteria:

1. Subjects meeting criteria for an eating disorder or an autistic spectrum disorder.
2. IQ below the mild mental retardation range (<60), based on verified records of cognitive testing performed within 2 years of enrollment. In event that suitable records of prior testing are unavailable, IQ will be estimated based on current classroom placement.
3. Significant medical and/or neurological illness, including seizure disorders, severe respiratory illness or cardiac conditions; cerebrovascular disease; hypo- or hypertension; immune, endocrine, renal, or hepatic dysfunction. The definition of such dysfunction will be derived from laboratory normal ranges, such that values lying outside those ranges would be considered abnormal.
4. Subjects taking antidepressants.
5. Active substance abuse/dependence based upon history and/or urine toxicology tests performed at screening.
6. Inability to have blood drawn at baseline, weekly, and termination visits.
7. Known allergy or hypersensitivity to metformin or its ingredients.
8. Recent history of suicidality, suicidal ideation, or suicide attempts.
9. Patients clinically unstable on current medication regimen.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
BMI | weekly

SECONDARY OUTCOMES:
MOSES | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Jean A Frazier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Medford, Massachusetts, United States